CLINICAL TRIAL: NCT00539136
Title: An Open-label, Single-dose, Non-randomized, Balanced Design Three-way Cross-over Study to Examine the Variability in Absorption of GSK561679 Using Gamma Scintigraphy, PillCam™ SB Capsule and the Acoustic Vest in Healthy Males Volunteers
Brief Title: A Study to Examine the Absorption of GSK561679 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CRS-110300
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Healthy Subjects
Keywords: GSK561679,; Pharmacokinetic,; healthy volunteers,; Gamma Scintigraphy,; PillCam™,; acoustic vest
MeSH Terms: interventions — NBI 77860; Solutions

INTERVENTIONS:
Drug: GSK561679 tablet or solution

SUMMARY:
This study will be conducted in healthy volunteers to investigate the absorption of GSK561679 using Gamma Scintigraphy, PillCam™ SB capsule and the acoustic vest.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18-55 years, inclusive.
* Healthy subjects, defined as individuals who are free from clinically significant illness or disease (including peptic ulcer disease and psychiatric illness) as determined by their medical and psychiatric history (including family), physical examination, laboratory studies, and other tests.
* Body weight >/= 50 kg (110 lbs) and BMI within the range 18.5-29.9 kg/m2 inclusive
* Demonstrates no evidence of active disease, physical or mental impairment.
* Self-administered Beck Depression Inventory II scale total score no greater than 9, and suicide question score of zero.
* Non-smoker (abstinence from smoking for at least 6 months before the start of the study).
* Normal electrocardiogram (subjects must have no clinically significant abnormalities on a 12-lead ECG).
* Agree to remain in the clinic for the time defined in the protocol.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* As a result of any of the medical interview, physical examination, evaluation of mental state and psychiatric history or screening investigations, the physician responsible considers the subject unfit for the study.
* History of clinically significant psychiatric illness.
* Any history of suicidal attempts or behavior.
* Any history of an endocrine disorder including, but not limited to, diabetes or disorders of the hypothalamus, pituitary, adrenal, or thyroid glands, or gonadal disorder or dysfunction of the reproductive organs.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, oesophageal reflux, irritable bowel syndrome or intestinal obstruction; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecystectomy) which would be expected to influence the absorption of drugs.
* History or presence of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* LFTs elevated >1.5 times above the reference range at pre-study screening that remain elevated with a repeat LFT (to be discussed with the sponsor, if necessary).
* Any other clinically significant laboratory abnormality.
* The subject has a screening ECG with values outside ranges specified in protocol.
* A semi-supine systolic blood pressure less than 90 mmHg or greater than 140 mmHg or a semi-supine diastolic blood pressure of less than 60 mmHg or greater than 90mmHg; or a radial pulse rate less than 40 bpm or more than 90 bpm.
* A positive pre-study HIV 1, Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of the start of the study. Subjects with a negative Hepatitis B, C and HIV test in last 3 months will not be required to repeat the tests.
* The subject has a positive pre-study urine drug/alcohol screen. .
* History of regular alcohol consumption averaging 21 drinks/week within 6 months of screening.
* Average daily caffeine intake equivalent to > 4 cups of coffee or > 6 cups of tea.
* Consumption of grapefruit juice or grapefruit within 14 days prior to the first dose of study medication.
* The subject is a vegetarian and/or has specific dietary requirements which would prevent them from eating the meals provided during the study.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* An unwillingness to use a condom/spermicide during sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until five half lives following administration of the last dose of study medication.
* An unwillingness to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until 84 days following administration of the last dose of study medication.
* The subject has received an investigational drug or participated in any other research trial within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug(whichever is longer) prior to the first dose of current study medication.
* Where participation in the study would result in donation of excess of 600 mL blood within a 56 day period.
* Radiation exposure, including that from the present study, exceeding a cumulative total effective dose equivalent of 10mSv over the last 3 years. Radiation exposure from previous clinical trials will be included, but clinical (therapeutic or diagnostic) radiation exposures will not be included.
* Radiation exposure from clinical trials, including that from present study, and from diagnostic X-rays, but excluding background radiation, exceeding a target organ (colon) dose of 50mSv (5 rems) from a single dose within the last 30 days or a cumulative dose of 150mSv (15 rems) in the last twelve (12) months. No subject whose occupation requires monitoring for radiation exposure will be enrolled in the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic scope of GSK561679 after application in a solution and in a new tablet formula per treatment phase Complete gastric emptying of radioactive marker after application of GSK561679 Complete tablet breakdown per treatment phase

SECONDARY OUTCOMES:
AUC(0-24h), AUC(0-t), AUC(0-∞) of GSK561679 after administration of GSK561679 in a solution (fasted) and in a new "optimized" tablet formulation (fasted and fed).
lambda_Z (and t1/2), tlag, Ka, the time to absorb the 25, 50 and 90% of the total absorbed dose
•Other pharmacokinetic parameters of GSK561679 per treatment phase •Safety and tolerability parameters, including adverse events, clinical laboratory,vital signs and 12-lead ECGs measured at each dosing period and throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Lexington, Kentucky, United States